CLINICAL TRIAL: NCT01039714
Title: Preoperative Vitamin D Levels as a Prognostic Factor for Postoperative Hypocalcemia and Hypoparathyroidism After Total Thyroidectomy
Brief Title: Vitamin D Levels and Postoperative Hypocalcemia After Total Thyroidectomy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Aristotle University Of Thessaloniki (Other)
Responsible Party: Third Surgical Clinic, AHEPA University Hospital, Third Surgical Clinic, AHEPA University Hospital
Other Study IDs: GXKVITD1
Record Dates: First submitted 2009-09-29; First posted 2009-12-25 (Estimated); Last update posted 2009-12-25 (Estimated); Status verified 2009-12

CONDITIONS: Hypocalcemia; Hypoparathyroidism; Vitamin D Deficiency; Thyroidectomy
Keywords: Hypocalcemia; Hypoparathyroidism; Vitamin D deficiency; Total thyroidectomy; calcium; PTH
MeSH Terms: conditions — Hypocalcemia; Hypoparathyroidism; Vitamin D Deficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Total Thyroidectomy

SUMMARY:
Hypocalcemia is one of the most frequent complications of total thyroidectomy, a procedure used for benign as well as malignant conditions of the thyroid gland. Postoperative hypocalcemia is usually caused by hypoparathyroidism. Vitamin D is implicated in calcium metabolism as it increases intestinal calcium transport and regulates parathormone production. Aim of the present study is to evaluate preoperative vitamin D levels as a prognostic factor for postoperative hypocalcemia and hypoparathyroidism.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is over 18 years old
2. Patient scheduled for total thyroidectomy
3. Patient signs and dates a written informed consent form (ICF) and indicates an understanding of the study procedures

Exclusion Criteria:

1. Primary hyperparathyroidism
2. Primary hypoparathyroidism
3. Chronic Renal Failure
4. Hypoalbuminemia
5. Neck irradiation
6. Systematic Diseases (e.g., infections)
7. Thyroid or parathyroid cancer
8. Osteoporosis
9. Drugs that influence calcium metabolism (vitamin D analogues, oral calcium supplements, biphosphonates, teriparatide, thiazide diuretics)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients subjected to total thyroidectomy in Third Surgical Clinic of AHEPA University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2009-12; Primary Completion 2010-04 (Estimated); Study Completion 2010-05 (Estimated)

PRIMARY OUTCOMES:
Impact of preoperative vitamin D levels on postoperative hypocalcemia after total thyroidectomy. | 24 hours postoperatively

SECONDARY OUTCOMES:
Impact of preoperative vitamin D levels on parathyroid function after total thyroidectomy. | 24 hours postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Spyros T Papavramidis, Prof, Study Director — Aristotle University Of Thessaloniki
Locations (1):
- AHEPA University Hospital Thessaloniki, Greece, Thessaloniki, Makedonia, Greece

REFERENCES:
- [Background] Erbil Y, Barbaros U, Temel B, Turkoglu U, Issever H, Bozbora A, Ozarmagan S, Tezelman S. The impact of age, vitamin D(3) level, and incidental parathyroidectomy on postoperative hypocalcemia after total or near total thyroidectomy. Am J Surg. 2009 Apr;197(4):439-46. doi: 10.1016/j.amjsurg.2008.01.032. PMID 19324110